CLINICAL TRIAL: NCT03274999
Title: Randomized, Controlled, Single-Center, Cross-Over Clinical Study to Evaluate Tear Characteristics Following Acute TrueTear™ Use
Brief Title: Clinical Study to Evaluate Tear Characteristics Following Acute TrueTear™ Use
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Based on interim review and decision to re-design the study.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OCUN-020
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Results first posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TrueTear™ Intranasal then Extranasal Application (Experimental): TrueTear™ device, intranasal (test) application, for approximately 3 minutes on Day 0 followed by TrueTear™ device, extranasal (control) application, for approximately 3 minutes on Day 14.
  Interventions: Device: TrueTear™ Application
- TrueTear™ Extranasal then Intranasal Application (Experimental): TrueTear™ device, extranasal (control) application, for approximately 3 minutes on Day 0 followed by TrueTear™ device, intranasal (test) application, for approximately 3 minutes on Day 14.
  Interventions: Device: TrueTear™ Application

INTERVENTIONS:
Device: TrueTear™ Application — Intranasal and extranasal application of TrueTear™ device for approximately 3 minutes at Day 0 and Day 14.

SUMMARY:
This study will evaluate the change in tear meniscus height (TMH) produced by intranasal stimulation with TrueTear™ compared with the same device applied extranasally (control).

ELIGIBILITY:
Inclusion Criteria:

* Baseline Ocular Surface Disease Index© (OSDI©) score of at least 23 with no more than three responses of "not applicable"
* In at least one eye, a baseline Schirmer test of ≤ 10 mm/5 minutes AND a cotton swab nasal stimulation Schirmer test of at least 7 mm higher in the same eye

Exclusion Criteria:

* Chronic or recurrent epistaxis, coagulation disorders or other conditions that may increase the risk of bleeding
* History of nasal or sinus surgery
* Vascularized polyp, deviated septum or severe nasal airway obstruction at the Screening visit
* Intraocular and extraocular surgery in either eye within three months of the Screening Visit or refractive surgery within twelve months of the Screening Visit
* Cardiac demand pacemaker, implanted defibrillator, or other active implanted metallic or active implanted electronic device in the head

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2017-11-09 (Actual); Study Completion 2017-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director, Study Director — Allergan, plc
Locations (1):
- Ocular Technology Group International, London, United Kingdom

REFERENCES:
- See also: For information to locate a study location near you, please visit AllerganClinicalTrials.com — http://AllerganClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (Day 0)
Arm/Group | TrueTear™ Intranasal Then Extranasal Application | TrueTear™ Extranasal Then Intranasal Application
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Intervention (Day 14)
Arm/Group | TrueTear™ Intranasal Then Extranasal Application | TrueTear™ Extranasal Then Intranasal Application
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received TrueTear™ either intranasally or extranasally.
Groups:
- All Study Participants: All participants randomized to receive TrueTear™ device either intranasally (test) or extranasally (control) on Days 0 and 14.
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All participants randomized to receive TrueTear ™ device either intranasally or extranasally on Days 0 and 14.
  years | 52.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Pre-application) in Tear Meniscus Height (TMH) at Eye Opening and Pre-Blink
Description: Tear meniscus height is defined as the mean height of the lower tear prism to the edge of the eye lid measured by the investigator using the Tear scope Plus in conjunction with a Topcon SL-D7 slit lamp biomicroscope and high-resolution digital video recording. Change from Baseline to time (T) T0 (immediately), T15, T30, T60, T120, T180, T240, T300, T360 minutes (mins) after application was reported. A negative change from Baseline (Pre-application) indicates improvement.
Time Frame: Pre-application (Day 0) to time (T) 0 (immediately), 15, 30, 60, 120, 180, 240, 300 and 360 minutes on Day 0 after application
Population: All participants who met the eligibility criteria, adhered to the protocol, and successfully completed the full study assessment were included in the per-protocol analysis.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- TrueTear™ Extranasal Application: TrueTear™ device, extranasal (control) application, for approximately 3 minutes on Day 0 or Day 14.
- TrueTear™ Intranasal Application: TrueTear™ device, intranasal (test) application, for approximately 3 minutes on Day 0 or Day 14.
Arm/Group | TrueTear™ Extranasal Application | TrueTear™ Intranasal Application
Number analyzed (Participants) | 10 | 10
mm
  Eye-opening,Pre-application,Day 0 | 0.312 (0.132) | 0.310 (0.143)
  Eye-opening,Change at T0 after application,Day 0 | 0.047 (0.205) | 0.105 (0.177)
  Eye-opening,Change at T15 after application,Day 0 | 0.010 (0.110) | 0.002 (0.096)
  Eye-opening,Change at T30 after application,Day 0 | -0.035 (0.118) | -0.003 (0.100)
  Eye-opening,Change at T60 after application,Day 0 | -0.018 (0.107) | -0.038 (0.092)
  Eye-opening,Change at T120 after application,Day 0 | -0.021 (0.138) | -0.039 (0.101)
  Eye-opening,Change at T180 after application,Day 0 | -0.049 (0.136) | -0.032 (0.103)
  Eye-opening,Change at T240 after application,Day 0 | -0.022 (0.125) | -0.033 (0.137)
  Eye-opening,Change at T300 after application,Day 0 | -0.055 (0.095) | -0.065 (0.110)
  Eye-opening,Change at T360 after application,Day 0 | -0.049 (0.111) | -0.060 (0.126)
  Pre-blink,Pre-application,Day 0 | 0.379 (0.152) | 0.350 (0.143)
  Pre-blink,Change at T0 after application,Day 0 | 0.067 (0.263) | 0.154 (0.231)
  Pre-blink,Change at T15 after application,Day 0 | 0.005 (0.143) | 0.027 (0.097)
  Pre-blink,Change at T30 after application,Day 0 | -0.040 (0.149) | 0.012 (0.105)
  Pre-blink,Change at T60 after application,Day 0 | -0.035 (0.159) | -0.008 (0.097)
  Pre-blink,Change at T120 after application,Day 0 | -0.050 (0.150) | -0.024 (0.097)
  Pre-blink,Change at T180 after application,Day 0 | -0.050 (0.153) | -0.039 (0.074)
  Pre-blink,Change at T240 after application,Day 0 | -0.018 (0.159) | -0.037 (0.132)
  Pre-blink,Change at T300 after application,Day 0 | -0.074 (0.133) | -0.070 (0.117)
  Pre-blink,Change at T360 after application,Day 0 | -0.054 (0.121) | -0.047 (0.129)
Statistical Analysis 1: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; The null hypothesis for the outcome measure is the difference in the change from the pre-application value at post-application time (T0) between the intranasal (test) and extranasal (control) applications are zero; Test type: Superiority; p = 0.156, t-test, 1 sided — Eye-opening, T0: P-value was calculated using 1-sided paired t-test
Statistical Analysis 2: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; The null hypothesis for the outcome measure is the difference in the change from the pre-application value at post-application time (T15) between the intranasal (test) and extranasal (control) applications are zero; Test type: Superiority; p = 0.395, t-test, 1 sided — Eye-opening, T15: P-value was calculated using 1-sided paired t-test
Statistical Analysis 3: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; The null hypothesis for the outcome measure is the difference in the change from the pre-application value at post-application time (T30) between the intranasal (test) and extranasal (control) applications are zero; Test type: Superiority; p = 0.114, t-test, 1 sided — Eye-opening, T30: P-value was calculated using 1-sided paired t-test
Statistical Analysis 4: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; The null hypothesis for the outcome measure is the difference in the change from the pre-application value at post-application time (T60) between the intranasal (test) and extranasal (control) applications are zero; Test type: Superiority; p = 0.211, t-test, 1 sided — Eye-opening, T60: P-value was calculated using 1-sided paired t-test
Statistical Analysis 5: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; The null hypothesis for the outcome measure is the difference in the change from the pre-application value at post-application time (T120) between the intranasal (test) and extranasal (control) applications are zero; Test type: Superiority; p = 0.332, t-test, 1 sided — Eye-opening, T120: P-value was calculated using 1-sided paired t-test
Statistical Analysis 6: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; The null hypothesis for the outcome measure is the difference in the change from the pre-application value at post-application time (T180) between the intranasal (test) and extranasal (control) applications are zero; Test type: Superiority; p = 0.318, t-test, 1 sided — Eye-opening, T180: P-value was calculated using 1-sided paired t-test
Statistical Analysis 7: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; The null hypothesis for the outcome measure is the difference in the change from the pre-application value at post-application time (T240) between the intranasal (test) and extranasal (control) applications are zero; Test type: Superiority; p = 0.375, t-test, 1 sided — Eye-opening, T240: P-value was calculated using 1-sided paired t-test
Statistical Analysis 8: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; The null hypothesis for the outcome measure is the difference in the change from the pre-application value at post-application time (T300) between the intranasal (test) and extranasal (control) applications are zero; Test type: Superiority; p = 0.352, t-test, 1 sided — Eye-opening, T300: P-value was calculated using 1-sided paired t-test
Statistical Analysis 9: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; The null hypothesis for the outcome measure is the difference in the change from the pre-application value at post-application time (T360) between the intranasal (test) and extranasal (control) applications are zero; Test type: Superiority; p = 0.312, t-test, 1 sided — Eye-opening, T360: P-value was calculated using 1-sided paired t-test
Statistical Analysis 10: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.134, t-test, 1 sided — Pre-blink, T0: P-value was calculated using 1-sided paired t-test
Statistical Analysis 11: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.315, t-test, 1 sided — Pre-blink, T15: P-value was calculated using 1-sided paired t-test
Statistical Analysis 12: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.071, t-test, 1 sided — Pre-blink, T30: P-value was calculated using 1-sided paired t-test
Statistical Analysis 13: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.260, t-test, 1 sided — Pre-blink, T60: P-value was calculated using 1-sided paired t-test
Statistical Analysis 14: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = 0.264, t-test, 1 sided — Pre-blink, T120: P-value was calculated using 1-sided paired t-test
Statistical Analysis 15: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 6]; Test type: Superiority; p = 0.381, t-test, 1 sided — Pre-blink, T180: P-value was calculated using 1-sided paired t-test
Statistical Analysis 16: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.249, t-test, 1 sided — Pre-blink, T240: P-value was calculated using 1-sided paired t-test
Statistical Analysis 17: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 8]; Test type: Superiority; p = 0.451, t-test, 1 sided — Pre-blink, T300: P-value was calculated using 1-sided paired t-test
Statistical Analysis 18: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 9]; Test type: Superiority; p = 0.393, t-test, 1 sided — Pre-blink, T360: P-value was calculated using 1-sided paired t-test

2. Primary Outcome: Change From Baseline (Pre-application) in Tear Lipid Layer Thickness at Eye Opening and Pre-Blink
Description: Lipid layer thickness is defined as the average thickness of the lipid layer calculated from the thickness of the various pattern weighted by the relative coverage of each pattern measured by the investigator using the Tearscope Plus in conjunction with a Topcon SL-D7 slit lamp biomicroscope and high-resolution digital video recording. Change from Baseline to T0 (immediately), T15, T30, T60, T120, T180, T240, T300, T360 mins after application was reported. A negative change from Baseline (Pre-application) indicates improvement .
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nm
Arm/Group | TrueTear™ Extranasal Application | TrueTear™ Intranasal Application
Number analyzed (Participants) | 10 | 10
nm
  Eye-opening,Pre-application,Day 0 | 41.090 (12.185) | 33.541 (9.848)
  Eye-opening,Change at T0 after application,Day 0 | 0.325 (19.890) | 25.255 (21.278)
  Eye-opening,Change at T15 after application,Day 0 | -2.527 (16.680) | 6.154 (9.924)
  Eye-opening,Change at T30 after application,Day 0 | -6.820 (14.292) | 6.944 (14.559)
  Eye-opening,Change at T60 after application,Day 0 | -2.542 (17.665) | 6.174 (13.224)
  Eye-opening,Change at T120 after application,Day 0 | -6.385 (16.423) | -0.310 (11.519)
  Eye-opening,Change at T180 after application,Day 0 | -2.766 (12.617) | 1.522 (9.387)
  Eye-opening,Change at T240 after application,Day 0 | -4.815 (16.918) | 2.212 (9.965)
  Eye-opening,Change at T300 after application,Day 0 | 0.481 (16.789) | 4.662 (12.366)
  Eye-opening,Change at T360 after application,Day 0 | -4.210 (14.388) | 1.320 (9.393)
  Pre-blink,Pre-application,Day 0 | 46.498 (19.880) | 45.330 (18.124)
  Pre-blink,Change at T0 after application,Day 0 | 3.907 (19.689) | 23.203 (24.003)
  Pre-blink,Change at T15 after application,Day 0 | -1.145 (17.824) | 4.018 (20.612)
  Pre-blink,Change at T30 after application,Day 0 | -3.662 (17.007) | -0.351 (19.049)
  Pre-blink,Change at T60 after application,Day 0 | 0.246 (20.592) | 2.990 (19.916)
  Pre-blink,Change at T120 after application,Day 0 | -4.684 (17.573) | -3.939 (13.767)
  Pre-blink,Change at T180 after application,Day 0 | -3.373 (14.149) | -4.464 (10.932)
  Pre-blink,Change at T240 after application,Day 0 | -1.033 (17.147) | -4.381 (14.947)
  Pre-blink,Change at T300 after application,Day 0 | 1.700 (20.157) | 1.725 (20.086)
  Pre-blink,Change at T360 after application,Day 0 | -3.730 (16.013) | -4.863 (13.992)
Statistical Analysis 1: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.006, t-test, 1 sided — Eye-opening, T0: P-value was calculated using 1-sided paired t-test
Statistical Analysis 2: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.063, t-test, 1 sided — Eye-opening, T15: P-value was calculated using 1-sided paired t-test
Statistical Analysis 3: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.005, t-test, 1 sided — Eye-opening, T30: P-value was calculated using 1-sided paired t-test
Statistical Analysis 4: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.089, t-test, 1 sided — Eye-opening, T60: P-value was calculated using 1-sided paired t-test
Statistical Analysis 5: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = 0.112, t-test, 1 sided — Eye-opening, T120: P-value was calculated using 1-sided paired t-test
Statistical Analysis 6: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 6]; Test type: Superiority; p = 0.16, t-test, 1 sided — Eye-opening, T180: P-value was calculated using 1-sided paired t-test
Statistical Analysis 7: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.077, t-test, 1 sided — Eye-opening, T240: P-value was calculated using 1-sided paired t-test
Statistical Analysis 8: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 8]; Test type: Superiority; p = 0.157, t-test, 1 sided — Eye-opening, T300: P-value was calculated using 1-sided paired t-test
Statistical Analysis 9: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 9]; Test type: Superiority; p = 0.111, t-test, 1 sided — Eye-opening, T360: P-value was calculated using 1-sided paired t-test
Statistical Analysis 10: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.040, t-test, 1 sided — Pre-blink, T0: P-value was calculated using 1-sided paired t-test
Statistical Analysis 11: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.241, t-test, 1 sided — Pre-blink, T15: P-value was calculated using 1-sided paired t-test
Statistical Analysis 12: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.284, t-test, 1 sided — Pre-blink, T30: P-value was calculated using 1-sided paired t-test
Statistical Analysis 13: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.313, t-test, 1 sided — Pre-blink, T60: P-value was calculated using 1-sided paired t-test
Statistical Analysis 14: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = 0.433, t-test, 1 sided — Pre-blink, T120: P-value was calculated using 1-sided paired t-test
Statistical Analysis 15: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 6]; Test type: Superiority; p = 0.406, t-test, 1 sided — Pre-blink, T180: P-value was calculated using 1-sided paired t-test
Statistical Analysis 16: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.318, t-test, 1 sided — Pre-blink, T240: P-value was calculated using 1-sided paired t-test
Statistical Analysis 17: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 8]; Test type: Superiority; p = 0.499, t-test, 1 sided — Pre-blink, T300: P-value was calculated using 1-sided paired t-test
Statistical Analysis 18: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 9]; Test type: Superiority; p = 0.390, t-test, 1 sided — Pre-blink, T360: P-value was calculated using 1-sided paired t-test

3. Primary Outcome: Change From Baseline (Pre-application) in Non-Invasive Tear Film Break-Up Time (NIBUT)
Description: Non-invasive break-up time is the time in seconds between eye opening and the appearance of the first visible break in the lipid layer of the pre-corneal tear film measured by the investigator using the Tearscope Plus in conjunction with a Topcon SL-D7 slit lamp biomicroscope and high-resolution digital video recording. Change from Baseline to T0 (immediately), T15, T30, T60, T120, T180, T240, T300, T360 mins after application was reported. A negative change from Baseline (Pre-application) indicates improvement.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | TrueTear™ Extranasal Application | TrueTear™ Intranasal Application
Number analyzed (Participants) | 10 | 10
seconds
  Pre-application, Day 0 | 18.211 (23.626) | 10.536 (8.458)
  Change at T0 after application, Day 0 | -2.668 (16.857) | 4.784 (13.738)
  Change at T15 after application, Day 0 | -2.489 (15.788) | 0.835 (8.258)
  Change at T30 after application, Day 0 | 3.561 (19.045) | -0.639 (7.272)
  Change at T60 after application, Day 0 | 6.951 (27.848) | -0.954 (9.171)
  Change at T120 after application, Day 0 | -0.128 (14.178) | 1.683 (7.172)
  Change at T180 after application, Day 0 | 4.911 (20.700) | -0.449 (6.029)
  Change at T240 after application, Day 0 | 1.525 (26.612) | -0.787 (9.026)
  Change at T300 after application, Day 0 | -0.387 (15.805) | -1.656 (5.560)
  Change at T360 after application, Day 0 | -1.509 (18.756) | -0.722 (8.369)
Statistical Analysis 1: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.053, t-test, 1 sided — T0: P-value was calculated using 1-sided paired t-test
Statistical Analysis 2: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.206, t-test, 1 sided — T15: P-value was calculated using 1-sided paired t-test
Statistical Analysis 3: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.221, t-test, 1 sided — T30: P-value was calculated using 1-sided paired t-test
Statistical Analysis 4: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.126, t-test, 1 sided — T60: P-value was calculated using 1-sided paired t-test
Statistical Analysis 5: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = 0.124, t-test, 1 sided — T120: P-value was calculated using 1-sided paired t-test
Statistical Analysis 6: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 6]; Test type: Superiority; p = 0.167, t-test, 1 sided — T180: P-value was calculated using 1-sided paired t-test
Statistical Analysis 7: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.377, t-test, 1 sided — T240: P-value was calculated using 1-sided paired t-test
Statistical Analysis 8: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 8]; Test type: Superiority; p = 0.397, t-test, 1 sided — T300: P-value was calculated using 1-sided paired t-test
Statistical Analysis 9: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 9]; Test type: Superiority; p = 0.441, t-test, 1 sided — T360: P-value was calculated using 1-sided paired t-test

4. Primary Outcome: Change From Pre-application in Protective Index (PI)
Description: The Protected Index (PI) corresponds to the percentage of the corneal surface that is not exposed to the atmosphere (i.e. fully covered by the tear film) over the full interblink period measured by the investigator using a Tear scope Plus in conjunction with a Topcon SL-D7 slit lamp biomicroscope and high-resolution digital video recording. Change from Baseline to T0 (immediately), T15, T30, T60, T120, T180, T240, T300, T360 mins after application was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of area covered by tear film
Arm/Group | TrueTear™ Extranasal Application | TrueTear™ Intranasal Application
Number analyzed (Participants) | 10 | 10
percentage of area covered by tear film
  Pre-application, Day 0 | 99.999 (0.004) | 98.797 (5.351)
  Change at T0 after application, Day 0 | -0.003 (0.015) | 1.200 (5.343)
  Change at T15 after application, Day 0 | 0.000 (0.001) | 1.198 (5.352)
  Change at T30 after application, Day 0 | -0.009 (0.036) | 1.196 (5.352)
  Change at T60 after application, Day 0 | 0.000 (0.007) | 1.196 (5.352)
  Change at T120 after application, Day 0 | 0.000 (0.002) | 1.179 (5.260)
  Change at T180 after application, Day 0 | 0.001 (0.004) | 1.193 (5.353)
  Change at T240 after application, Day 0 | -0.005 (0.020) | 1.196 (5.352)
  Change at T300 after application, Day 0 | -0.004 (0.017) | 1.196 (5.352)
  Change at T360 after application, Day 0 | 0.000 (0.003) | 1.198 (5.352)
Statistical Analysis 1: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.034, t-test, 1 sided — T0: P-value was calculated using 1-sided paired t-test
Statistical Analysis 2: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.143, t-test, 1 sided — T15: P-value was calculated using 1-sided paired t-test
Statistical Analysis 3: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.328, t-test, 1 sided — T30: P-value was calculated using 1-sided paired t-test
Statistical Analysis 4: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.250, t-test, 1 sided — T60: P-value was calculated using 1-sided paired t-test
Statistical Analysis 5: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = 0.090, t-test, 1 sided — T120: P-value was calculated using 1-sided paired t-test
Statistical Analysis 6: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 6]; Test type: Superiority; p = 0.328, t-test, 1 sided — T180: P-value was calculated using 1-sided paired t-test
Statistical Analysis 7: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.055, t-test, 1 sided — T240: P-value was calculated using 1-sided paired t-test
Statistical Analysis 8: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 8]; Test type: Superiority; p = 0.090, t-test, 1 sided — T300: P-value was calculated using 1-sided paired t-test
Statistical Analysis 9: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 9]; Test type: Superiority; p = 0.233, t-test, 1 sided — T360: P-value was calculated using 1-sided paired t-test

5. Primary Outcome: Change From Pre-application in Exposed Area (EA)
Description: Exposed Area is defined as the percentage of the observed area not covered by the tear film at the time of the blink hence exposed to the atmosphere measured by the investigator using a Tear scope Plus in conjunction with a Topcon SL-D7 slit lamp biomicroscope and high-resolution digital video recording. Change from Baseline to T0 (immediately), T15, T30, T60, T120, T180, T240, T300, T360 mins after application was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage area not covered by tear film
Arm/Group | TrueTear™ Extranasal Application | TrueTear™ Intranasal Application
Number analyzed (Participants) | 10 | 10
percentage area not covered by tear film
  Pre-application, Day 0 | 0.005 (0.022) | 0.022 (0.057)
  Change at T0 after application, Day 0 | 0.014 (0.077) | -0.014 (0.035)
  Change at T15 after application, Day 0 | -0.002 (0.010) | -0.006 (0.046)
  Change at T30 after application, Day 0 | 0.033 (0.140) | -0.008 (0.051)
  Change at T60 after application, Day 0 | -0.001 (0.029) | 0.001 (0.088)
  Change at T120 after application, Day 0 | -0.004 (0.016) | 0.028 (0.145)
  Change at T180 after application, Day 0 | -0.005 (0.022) | 0.011 (0.086)
  Change at T240 after application, Day 0 | 0.012 (0.040) | -0.008 (0.091)
  Change at T300 after application, Day 0 | 0.005 (0.022) | -0.002 (0.052)
  Change at T360 after application, Day 0 | -0.001 (0.018) | -0.006 (0.051)
Statistical Analysis 1: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.072, t-test, 1 sided — T0: P-value was calculated using 1-sided paired t-test
Statistical Analysis 2: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.297, t-test, 1 sided — T15: P-value was calculated using 1-sided paired t-test
Statistical Analysis 3: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.328, t-test, 1 sided — T30: P-value was calculated using 1-sided paired t-test
Statistical Analysis 4: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.447, t-test, 1 sided — T60: P-value was calculated using 1-sided paired t-test
Statistical Analysis 5: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 5]; Test type: Superiority; p = 0.328, t-test, 1 sided — T120: P-value was calculated using 1-sided paired t-test
Statistical Analysis 6: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 6]; Test type: Superiority; p = 0.090, t-test, 1 sided — T180: P-value was calculated using 1-sided paired t-test
Statistical Analysis 7: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.055, t-test, 1 sided — T240: P-value was calculated using 1-sided paired t-test
Statistical Analysis 8: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 8]; Test type: Superiority; p = 0.090, t-test, 1 sided — T300: P-value was calculated using 1-sided paired t-test
Statistical Analysis 9: Comparison: TrueTear™ Extranasal Application vs TrueTear™ Intranasal Application; [analysis description as in outcome 1, analysis 9]; Test type: Superiority; p = 0.500, t-test, 1 sided — T360: P-value was calculated using 1-sided paired t-test

ADVERSE EVENTS:
Time Frame: Day 0 up to Day 14
Description: Safety population included all participants that initiated at least one application.
Arm/Group | TrueTear™ Extranasal Application | TrueTear™ Intranasal Application
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT03274999/Prot_SAP_000.pdf